CLINICAL TRIAL: NCT01365728
Title: A Prospective Randomized Comparison of Fellow Eyes Undergoing LASIK With the Intralase FS 60 Versus the Intralase IFS
Brief Title: An Outcomes Study Comparing the Intralase FS 60 to the Intralase iFS When Performing LASIK Surgery for Nearsightedness
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Other Study IDs: SU-05212011-7804; Stanford IRB Protocol # 21250
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Myopia; Astigmatism
Keywords: Femtosecond Laser; FS60; iFS; Intralase; Wavefront-guided LASIK; IntraLASIK; LASIK; Myopia; Nearsightedness
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: LASIK with the iFS femtosecond laser — Patients will undergo bilateral simultaneous LASIK surgery for myopia. One eye will have a LASIK flap created with the Intralase FS60 and the fellow eye will have a LASIK flap created with the Intralase iFS. Both eyes will undergo wavefront-guided LASIK surgery with the Visx CustomVue excimer laser.

SUMMARY:
The purpose of the study is to compare the results of LASIK surgery when using two versions of a femtosecond laser in patients with nearsightedness with and without astigmatism.

DETAILED DESCRIPTION:
The patients will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the patient from the study, then we will inform the patient and make an appropriate referral. if the patient is deemed appropriate for the study after a comprehensive examination included computerized videokeratography, then they can be enrolled. The patient will undergo bilateral simultaneous eye surgery. Which eye is treated with the Intralase FS 60 and which eye is treated with Intralase IFS will be randomized so there is a 50% chance for either eye to receive one treatment. The patients will be seen on the day of surgery, post op day one, one month, three months, six months and one year. The patient will receive topical antibiotics in each eye for one week following the procedure. The patient will receive pred forte 1% ophthalmic drops for one week after treatment. The patient will also receive vigamox ophthalmic drops for four days after treatment. All of this is within the usual and customary standard of care for the treatment of patients undergoing LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -0.25 diopters and -7.00 diopters with or without astigmatism of up to 3.00 diopters.

Exclusion Criteria:

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with ectactic eye disorders.
* Patients with autoimmune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects age 21 and older with healthy eyes. Nearsightedness between -0.25 diopters and -7.00 diopters with or without astigmatism of up to 3.00 diopters.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in Best Spectacle Corrected Visual Acuity | One year
Changes in 5% low contrast best corrected visual acuity | One year
Changes in corneal sensation | One year
Uncorrected Visual Acuity | One year
Stability of refractive outcome | One year
Changes in 25% low contrast best corrected visual acuity | One year

SECONDARY OUTCOMES:
Subjective Questionnaire | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States